CLINICAL TRIAL: NCT03964012
Title: Phase 3, Observer-blind, Randomized, Active Controlled Trial to Assess the Safety of an Investigational Meningococcal Serogroups ACYWX Conjugate Vaccine (NmCV-5) and Compare Its Immunogenicity to a Licensed Meningococcal Serogroups ACYW Conjugate Vaccine (Menactra®), in Healthy Subjects 2 to 29 Years of Age
Brief Title: Study to Assess Immunegnicity & Safety of Pentavalent Meningococcal Vaccine (NmCV-5)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACYWX-03; CVIA 071 (Other: PATH)
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2020-05

CONDITIONS: Meningococcal Meningitis
Keywords: Neisseria meningitidis; conjugate meningococcal vaccine; Meningococcal serogroup X
MeSH Terms: conditions — Meningitis, Meningococcal | interventions — NmCV-5 vaccine; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NmCV-5 (Experimental): Subjects in this arm will receive polyvalent conjugated vaccine against meningococcal serogroups A,C,Y,W & X.
  A single dose of 0.5 mL will be administered intramuscularly.
  Interventions: Biological: NmCV-5
- Menactra (Active Comparator): Subjects in this arm will licensed quadrivalent conjugated vaccine against meningococcal serogroups A,C,Y, & W viz. Menactra.
  A single dose of 0.5 mL will be administered intramuscularly.
  Interventions: Biological: Menactra

INTERVENTIONS:
Biological: NmCV-5 — Polyvalent conjugate meningococcal vaccine against serogroups A,C,Y,W&X (NmCV-5) is available as lyophilised powder of polysaccharide antigens A&X conjugated to tetanus toxoid and C,Y&W conjugated to C reactive material (CRM) protein. The diluent is Normal Saline. Each antigen content is 5 micrograms per 0.5 mL dose of vaccine.
  Other Names: MenACYWX
  Arms: NmCV-5
Biological: Menactra — Menactra is available as ready to use solution containing polysaccharide antigens A,C,Y&WX conjugated to diphtheria toxoid. Each antigen content is 4 micrograms per 0.5 mL dose of vaccine
  Other Names: MenACYW-D
  Arms: Menactra

SUMMARY:
This observer-blind, randomized, active controlled trial will be conducted among 2-29 year olds in two sites (Mali and The Gambia). The objectives of the study are to assess and compare the immunogenicity and safety of NmCV-5 with that of Menactra.

A total of 1800 eligible participants (who or their parents/guardians have given written informed consent) will be randomised 2:1 (NmCV-5: Menactra) in each of the three age strata 18-29 years, 11-17 years & 2-10 years (400 NmCV-5 recipients & 200 Menactra recipients in each age strata).

Each subject will receive a single dose of study vaccine and will be followed up for 6 months post vaccination during which solicited reactions (for seven days), unsolicited AEs (28 days) and SAEs (until the end of study i.e. 168 days after vaccination) will be collected. A blood sample will be collected at baseline (pre-vaccination) and at day 28 post-vaccination for immunogenicity assessment by a Serum Bactericidal Activity assay using rabbit complement (rSBA).

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female 2 through 29 years of age, inclusive, at the time of study IP administration.
2. Written informed consent obtained from subjects at least 18 years of age or from their parent/guardian for subjects less than 18 years of age with additional subject assent obtained as appropriate for participating community (i.e. subjects at least 13 years of age in Mali or at least 12 years of age in The Gambia).
3. Subject or parent/guardian with subject reside in study site area and are able and willing to adhere to all protocol visits and procedures.
4. Female subjects of childbearing potential must have practiced adequate contraception for 28 days prior to study IP administration and agree to continue adequate contraception until completion of their Day 29 visit.
5. Female subjects of childbearing potential must have a negative pregnancy test within 24 hours prior to study IP administration

Exclusion Criteria:

1. Acute illness, at the time of study IP administration (once acute illness is resolved, if appropriate, as per investigator assessment, subject may be re-revaluated for eligibility).
2. Recorded fever (for eligibility purpose defined as a body temperature greater than 37.5°C) within 3 days prior to study IP administration (once fever/acute illness is resolved, if appropriate, as per investigator assessment, subject may be re-revaluated for eligibility).
3. Previous immunization with a Neisseria meningitidis vaccine other than MenAfriVac® during the previous five years.
4. Current or previous, confirmed disease caused by Neisseria meningitidis.
5. Household contact with or intimate exposure to an individual with any laboratory confirmed Neisseria meningitidis infection within 90 days prior to study IP administration.
6. Known hypersensitivity to any component of the study IPs (i.e., NmCV-5 or Menactra®).
7. History of significant hypersensitivity reactions to any previous vaccine.
8. Administration of any vaccine other than study IPs within 28 days prior to study IP administration or planned administration prior to completion of the study Day 29 visit.
9. Administration of any investigational drug within 30 days prior to study IP administration or planned administration during the study period.
10. Unwilling to avoid (or their child to avoid, if the subject) the ingestion of herbal or other traditional medications during the study period.
11. Administration of immunoglobulin or any blood product within 90 days prior to study IP administration or planned administration during the study period.
12. Administration of immunosuppressants or other immune modifying agents within 90 days prior to study IP administration
13. Administration of systemic antibiotic treatment within 3 days prior to study IP administration.
14. Any history of or evidence for chronic clinically significant (as per investigator assessment) disorder or disease (including, but not limited to, immunodeficiency, autoimmunity, malnutrition, congenital abnormality, bleeding disorder, and pulmonary, cardiovascular, metabolic, neurologic, renal, or hepatic disease).
15. Any history of human immunodeficiency virus, chronic hepatitis B or chronic hepatitis C infections.
16. History of meningitis, seizures, Guillain-Barré syndrome (GBS), or other neurological disorders.
17. History of or family history of congenital or hereditary immunodeficiency.
18. Any condition that in the opinion of the investigator might compromise the safety or well-being of the subject or compromise adherence to protocol procedures or interfere with planned safety and immunogenicity assessments.
19. Pregnancy
20. Previous inclusion in the study of five immediate family members (i.e., biological father, mother, subject, and brothers and sisters may be included up to a maximum of five members from the same immediate family).

Ages: 2 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1800 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-02-23 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Seroresponse | 28 Days post vaccination
  Percentage of subjects with seroresponse, measured by rabbit complement serum bactericidal activity (rSBA) against serogroups A, C, Y, W and X. [Seroresponse is defined as a post-immunization (Day 29) rSBA titer of 32 or greater if the subject's pre-immunization (Day 1) rSBA titer was < 8; or a ≥ four-fold increase over baseline at Day 29 post-immunization if the subject's pre-immunization (Day 1) rSBA titer was ≥ 8].
Geometric mean titres | 28 Days post vaccination
  Geometric mean titers (GMTs) measured by rSBA against serogroups A, C, Y, W and X on Day 29

SECONDARY OUTCOMES:
Solicited adverse events | 7 days post vaccination
  Solicited AEs for 7 days following vaccination
Unsolicited adverse events | 28 days post vaccination
  Unsolicited AEs for 28 days following vaccination
Serious adverse events (SAEs) | 6 months post vaccination
  SAEs for 6 months following vaccination
Seroprotective rSBA titres | 28 days post vaccination
  Percentage of subjects with rSBA titer of ≥ 8 against serogroups A, C, Y, W, and X at Day 1 and Day 29
Long term protective rSBA titres | 28 days post vaccination
  Percentage of subjects with rSBA titer of ≥ 128 against serogroups A, C, Y, W, and X at Day 1 and Day 29

CONTACTS AND LOCATIONS:
Locations (2):
- Centre pour le Développement des Vaccins du Mali, ex-Institut Marchoux, Ministry of Health, BP251, Bamako, Mali
- Medical Research Council Unit The Gambia at the London School of Hygiene & Tropical Medicine, Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen WH, Neuzil KM, Boyce CR, Pasetti MF, Reymann MK, Martellet L, Hosken N, LaForce FM, Dhere RM, Pisal SS, Chaudhari A, Kulkarni PS, Borrow R, Findlow H, Brown V, McDonough ML, Dally L, Alderson MR. Safety and immunogenicity of a pentavalent meningococcal conjugate vaccine containing serogroups A, C, Y, W, and X in healthy adults: a phase 1, single-centre, double-blind, randomised, controlled study. Lancet Infect Dis. 2018 Oct;18(10):1088-1096. doi: 10.1016/S1473-3099(18)30400-6. Epub 2018 Aug 14. PMID 30120069
- [Derived] Castilla J, Cenoz MG, Barricarte A. Meningococcal Group B Vaccine (4CMenB) in Children. Reply. N Engl J Med. 2023 Jun 1;388(22):2109. doi: 10.1056/NEJMc2303518. No abstract available. PMID 37256992
- [Derived] Lopez-Lacort M, Munoz-Quiles C, Orrico-Sanchez A. Meningococcal Group B Vaccine (4CMenB) in Children. N Engl J Med. 2023 Jun 1;388(22):2109. doi: 10.1056/NEJMc2303518. No abstract available. PMID 37256991
- [Derived] Haidara FC, Umesi A, Sow SO, Ochoge M, Diallo F, Imam A, Traore Y, Affleck L, Doumbia MF, Daffeh B, Kodio M, Wariri O, Traore A, Jallow E, Kampmann B, Kapse D, Kulkarni PS, Mallya A, Goel S, Sharma P, Sarma AD, Avalaskar N, LaForce FM, Alderson MR, Naficy A, Lamola S, Tang Y, Martellet L, Hosken N, Simeonidis E, Welsch JA, Tapia MD, Clarke E. Meningococcal ACWYX Conjugate Vaccine in 2-to-29-Year-Olds in Mali and Gambia. N Engl J Med. 2023 May 25;388(21):1942-1955. doi: 10.1056/NEJMoa2214924. PMID 37224196